CLINICAL TRIAL: NCT06783946
Title: The Effect of Meditation on Anxiety and Pain of Patients Undergoing Ureteroscopy for Kidney Stones: A Pilot Randomized Study
Brief Title: Meditation Effects on Discomfort, Pain InTerference, and AnxieTy After urEteroscopy
Acronym: MEDITATE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-022475
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stone; Pain, Postoperative; Anxiety Postoperative
Keywords: Meditation; Post-Operative Pain; Ureteroscopy; Kidney Stones
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Block randomization, stratified by site, will be used to randomize participants into the treatment or control arms. Those in the treatment group will be taught a meditation intervention to be performed daily from 2-4 weeks before scheduled surgery date (whichever is the maximum length of time) to 2 weeks post-operatively. Participants will complete questionnaires to assess pain, anxiety, and depression at enrollment (day 0), post-operative days 3, 14, and 30. Participant feedback to assess experiences with the meditation intervention will be assessed within 1 month after completion of the final questionnaires.
Who Masked: Care Provider
Masking Description: Urologic surgeons who will be performing the ureteroscopy will be masked to the group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation (Experimental): In the intervention group, a meditation intervention will be implemented pre- and post-operatively. The meditation technique will be comprised of breathing techniques, full body relaxation, color meditation, visualization, and positive affirmations. A physician researcher trained in teaching meditation will conduct virtual meditation sessions with patients enrolled in the study. Participants will practice a daily 20-minute meditation for 2-4 weeks before scheduled surgery (whichever is the maximum length of time from enrollment) to 2 weeks post-operatively using the provided audio guided meditation recordings. Participants will also log adherence to meditation via daily questionnaires. They will receive standard pre-operative counseling and post-operative medications at the discretion of their urologist.
  Interventions: Behavioral: Meditation
- Usual Care (No Intervention): Those in the control or usual care arm will complete the same questionnaires at baseline and at post-operative days 3, 14, and 30. They will receive standard pre-operative counseling and post-operative medications at the discretion of their urologist.

INTERVENTIONS:
Behavioral: Meditation — The meditation technique will be comprised of breathing techniques, full body relaxation, color meditation, visualization, and positive affirmations. A physician researcher trained in teaching meditation will conduct virtual meditation sessions with patients enrolled in the study. Participants will practice a daily 20-minute meditation for 2-4 weeks before scheduled surgery (whichever is the maximum length of time from enrollment) to 2 weeks post-operatively using the provided audio guided meditation recordings. Participants will also log completion of daily meditation practice electronically.
  Arms: Meditation

SUMMARY:
The goal of this pilot clinical trial is to learn whether meditation can help improve recovery in children and adults having surgery for kidney stones. The main questions it aims to answer are:

* Does meditation around the time of surgery improve pain and anxiety in patients undergoing kidney stone surgery (ureteroscopy)?
* Is a meditation program around the time of surgery feasible for patients having kidney stone surgery (ureteroscopy)?

Participants will be randomly assigned to the meditation group and the control group to understand how meditation affects recovery after surgery. Participants will be asked to:

* Complete a health history form
* Complete questionnaires about pain and mood before surgery and certain days after surgery
* Those in the meditation group will learn and practice a daily 20-minute meditation for 2-4 weeks before surgery and 2 weeks after surgery
* Those in the meditation group will be asked to provide feedback of the meditation program after completing the last questionnaire

DETAILED DESCRIPTION:
Context:

Pain is common after surgery to remove urinary stones, and current options for post-operative pain management are limited. Pre-operative anxiety is a well-known clinical entity that is associated with a higher risk of post-operative pain. Meditation is an ancient discipline that has been used for a wide range of presumed benefits including improving pain and anxiety. Meditation has been studied in a variety of clinical settings, but its effects have not been assessed among patients having ureteroscopy to remove kidney and/or ureteral stones.

Objectives:

To determine the effect of a peri-operative meditation intervention on physical and emotional health in adolescent and adult patients undergoing elective unilateral ureteroscopy for unilateral renal or ureteral stones.

To determine the feasibility of implementing a perioperative meditation intervention in patients undergoing elective unilateral ureteroscopy for ureteral or renal stones

Study Design:

Pilot randomized controlled trial

Setting/Participants:

This study will recruit 50 patients aged 12 years or older at the Children's Hospital of Philadelphia and University of Pennsylvania, who will be undergoing elective unilateral ureteroscopy for unilateral renal or ureteral stones with or without stent placement. Participants will be randomized to the meditation intervention or usual care treatment arms.

Intervention: Participants will be randomized to the intervention (meditation) or control groups. Participants will learn and practice a daily 20-minute meditation for 2-4 weeks before scheduled surgery (whichever is the maximum length of time from enrollment) to 2 weeks post-operatively using the provided audio guide.

The Patient-Reported Outcomes Measurement Information System (PROMIS) instruments in the domains of Pain Intensity, Pain Interference, Anxiety, and Depression will be utilized. Patients will complete the questionnaire at the time of enrollment, and at post-operative days 3, 14, and 30. General information, health history, and kidney stone related events will be assessed from the medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 12 years and older
2. Diagnosis of unilateral or bilateral ureteral or renal stones
3. Scheduled to undergo elective unilateral ureteroscopy for renal or ureteral stones in 2 or more weeks from initial clinic visit
4. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Participants <12 years of age
2. Subjects undergoing any other type of stone procedure (i.e. bilateral ureteroscopy, percutaneous nephrolithotomy, ESWL, staged ureteroscopy)
3. Patients who are pre-stented at the initial clinic visit
4. Non-English speaking participants
5. Participants without functional e-mail address or phone
6. Participants unable to use a computer/tablet independently
7. Participants who will be undergoing ureteroscopy in less than 2 weeks from initial clinic visit
8. Patients who are non-verbal or with cognitive delay that may impair ability to learn and adhere to intervention
9. Patients with neurologic comorbidities that may alter sensation (eg. spinal cord injuries)
10. Parents/guardians or subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 3 (Pain Intensity) | Pre-operative baseline to post-operative day 3
  The primary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 3 in the domains of pain intensity, pain interference, anxiety, and depression.
  Four PROMIS questionnaires will be utilized, one for each domain. Questionnaires will be administered electronically with computerized adaptive testing (CAT). With CAT participants' responses guide the system's choice of subsequent items from the question bank; therefore, there is not a set number of questions per respondent. Each questionnaire will typically consist of 4-12 items and can be completed under 1 minute.
  Each questionnaire results in a standardized T-Score, in which 50 is the mean score for a general reference population, and 10 is the standard deviation. A higher PROMIS T-score represents more of the concept being measures (e.g. worse anxiety or pain intensity).
  Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain.
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 3 (Pain Interference) | Pre-operative baseline to post-operative day 3
  The primary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 3 in the domains of pain intensity, pain interference, anxiety, and depression.
  Four PROMIS questionnaires will be utilized, one for each domain. Questionnaires will be administered electronically with computerized adaptive testing (CAT). With CAT participants' responses guide the system's choice of subsequent items from the question bank; therefore, there is not a set number of questions per respondent. Each questionnaire will typically consist of 4-12 items and can be completed under 1 minute.
  Each questionnaire results in a standardized T-Score, in which 50 is the mean score for a general reference population, and 10 is the standard deviation. A higher PROMIS T-score represents more of the concept being measures (e.g. worse anxiety or pain intensity).
  Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain.
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 3 (Anxiety) | Pre-operative baseline to post-operative day 3
  The primary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 3 in the domains of pain intensity, pain interference, anxiety, and depression.
  Four PROMIS questionnaires will be utilized, one for each domain. Questionnaires will be administered electronically with computerized adaptive testing (CAT). With CAT participants' responses guide the system's choice of subsequent items from the question bank; therefore, there is not a set number of questions per respondent. Each questionnaire will typically consist of 4-12 items and can be completed under 1 minute.
  Each questionnaire results in a standardized T-Score, in which 50 is the mean score for a general reference population, and 10 is the standard deviation. A higher PROMIS T-score represents more of the concept being measures (e.g. worse anxiety or pain intensity).
  Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain.
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 3 (Depression) | Pre-operative baseline to post-operative day 3
  The primary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 3 in the domains of pain intensity, pain interference, anxiety, and depression.
  Four PROMIS questionnaires will be utilized, one for each domain. Questionnaires will be administered electronically with computerized adaptive testing (CAT). With CAT participants' responses guide the system's choice of subsequent items from the question bank; therefore, there is not a set number of questions per respondent. Each questionnaire will typically consist of 4-12 items and can be completed under 1 minute.
  Each questionnaire results in a standardized T-Score, in which 50 is the mean score for a general reference population, and 10 is the standard deviation. A higher PROMIS T-score represents more of the concept being measures (e.g. worse anxiety or pain intensity).
  Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain.

SECONDARY OUTCOMES:
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 30 (Pain Intensity) | Pre-operative baseline to 1 month post-operatively
  The secondary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 30 in the domains of pain intensity, pain interference, anxiety, and depression. Four PROMIS questionnaires will be used, one per domain. They will be administered electronically with computerized adaptive testing, where responses guide subsequent item selection from the question bank. Thus, there is not a set number of questions per respondent. Each questionnaire typically consists of 4-12 items and can be completed under 1 minute. Each questionnaire results in a standardized T-Score (50 is the mean for a general reference population, 10 is the standard deviation). A higher T-score represents more of the concept being measures (e.g. worse pain intensity). Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain. The trend of mean PROMIS T-Scores over the peri-operative period in both groups will be assessed.
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 30 (Pain Interference) | Pre-operative baseline to 1 month post-operatively
  The secondary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 30 in the domains of pain intensity, pain interference, anxiety, and depression. Four PROMIS questionnaires will be used, one per domain. They will be administered electronically with computerized adaptive testing, where responses guide subsequent item selection from the question bank. Thus, there is not a set number of questions per respondent. Each questionnaire typically consists of 4-12 items and can be completed under 1 minute. Each questionnaire results in a standardized T-Score (50 is the mean for a general reference population, 10 is the standard deviation). A higher T-score represents more of the concept being measures (e.g. worse pain intensity). Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain. The trend of mean PROMIS T-Scores over the peri-operative period in both groups will be assessed.
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 30 (Anxiety) | Pre-operative baseline to 1 month post-operatively
  The secondary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 30 in the domains of pain intensity, pain interference, anxiety, and depression. Four PROMIS questionnaires will be used, one per domain. They will be administered electronically with computerized adaptive testing, where responses guide subsequent item selection from the question bank. Thus, there is not a set number of questions per respondent. Each questionnaire typically consists of 4-12 items and can be completed under 1 minute. Each questionnaire results in a standardized T-Score (50 is the mean for a general reference population, 10 is the standard deviation). A higher T-score represents more of the concept being measures (e.g. worse pain intensity). Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain. The trend of mean PROMIS T-Scores over the peri-operative period in both groups will be assessed.
Change in PROMIS Scores from Pre-Operatively to Post-Operative Day 30 (Depression) | Pre-operative baseline to 1 month post-operatively
  The secondary outcome is the change in PROMIS T-scores from pre-operatively to post-operative day 30 in the domains of pain intensity, pain interference, anxiety, and depression. Four PROMIS questionnaires will be used, one per domain. They will be administered electronically with computerized adaptive testing, where responses guide subsequent item selection from the question bank. Thus, there is not a set number of questions per respondent. Each questionnaire typically consists of 4-12 items and can be completed under 1 minute. Each questionnaire results in a standardized T-Score (50 is the mean for a general reference population, 10 is the standard deviation). A higher T-score represents more of the concept being measures (e.g. worse pain intensity). Questionnaires will be administered at baseline and post-operative days 3, 14, 30 with separate T-scores for each time point and domain. The trend of mean PROMIS T-Scores over the peri-operative period in both groups will be assessed.
Feasibility Outcome: Monthly Proportion of Enrolled to Eligible Participants | Pre-operative baseline to 1 month post-operatively
  Measures of feasibility of implementation of a perioperative meditation intervention in patients undergoing elective unilateral ureteroscopy for ureteral or renal stones. This will include evaluating the proportion of enrolled to eligible participants per month, reported using descriptive statistics. Monthly enrollment proportions will be presented, along with the overall mean and range for the entire study enrollment period.
Feasibility Outcome: Completion of Questionnaires | Pre-operative baseline to 1 month post-operatively
  Measures of feasibility for implementing a perioperative meditation intervention in patients undergoing elective unilateral ureteroscopy for ureteral or renal stones will be assessed. This includes evaluating the proportion of PROMIS questionnaires completed at each time point, reported as the mean proportion of completed questionnaires to total eligible questionnaires, separated by group and by time point (baseline, post-operative days 3, 14, and 30).
Feasibility Outcome: Meditation Adherence | Pre-operative baseline to 1 month post-operatively
  Measures of feasibility for implementing a perioperative meditation intervention in patients undergoing elective unilateral ureteroscopy for ureteral or renal stones will include evaluating meditation session adherence. Participants in the intervention arm will complete daily online logs indicating whether meditation was performed (yes/no). Adherence will be calculated as the proportion of meditation days marked "yes" to the total eligible meditation days. Results will be summarized using descriptive statistics, including mean, median, and mode.
Number of Participants Who Sought Unplanned Medical Attention | Pre-operative baseline to 1 month post-operatively
  The number of participants seeking unplanned medical attention within 1 month post-operatively (including emergency department visits, unplanned office visits, unplanned surgical re-treatment, and phone calls) will be assessed through chart review and health care utilization questionnaires on post-operative days 14 and 30. Results will be reported as the mean number of unplanned medical events per participant.
Medication usage | From surgery to post-operative day 30
  A 2-item questionnaire will be administered to assess post-operative medication usage at post-operative days 3, 14, and 30. This will include:
  1. Has the participant taken any of these medications since surgery? Please select all medications at apply.
  2. Which of these medications is the participant currently taking? Please select all that apply.
  Medication options include a variety of over the counter and prescription medications typically prescribed after stone surgery.
  Number and type of medications taken will be assessed at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory E Tasian, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No